CLINICAL TRIAL: NCT00357227
Title: Atrial Fibrillation and the Risk for Neurological Complications
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Other Study IDs: 01 GI 0204
Record Dates: First submitted 2006-07-25; First posted 2006-07-27 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Stroke; Vascular Dementia; Mild Cognitive Impairment
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Dementia, Vascular; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
B8: Atrial fibrillation and the risk of neurological complications

Twenty-five thousand acute strokes are caused by atrial fibrillation every year. But even more frequent than symptomatic strokes are silent infarctions of the brain. Silent strokes remain undetected in most cases, but cumulate over time and progressively impair cognition. The impact of atrial fibrillation on subacute brain infarctions is not yet known. Moreover, it has not been elucidated so far how effective different therapeutic strategies in the treatment of atrial fibrillation prevent cognitive impairment. Thus, this study aims at evaluating the influence of different types of atrial fibrillation on silent strokes and the related impairment in cognitive functions. Other risk factors and cardiovascular diseases that are known to provoke the development of strokes will be assessed as well. So, it will be possible to isolate the contribution of atrial fibrillation to silent strokes and related cognitive impairment in segregation to other relevant factors. AF patients and controls will be examined twice in two years in order to evaluate the role of atrial fibrillation and differential therapeutic interventions with regard to the progression of silent strokes and cognitive impairment in a within subject-design.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of permanent, paroxysmal or episodic atrial fibrillation in the past or at present

Exclusion Criteria:

* Pacemaker
* Metal implants
* History of acute stroke
* Diagnosis of vascular or degenerative dementia
* History of brain tumors
* History of severe brain injury
* History of psychiatric disorders
* Pregnancy

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2004-01

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Knecht, Prof., Principal Investigator — University Hospital Münster, Department of Neurology
Locations (1):
- University Hospital Münster, Dept. of Neurology, Münster, North Rhine-Westphalia, Germany